CLINICAL TRIAL: NCT05782933
Title: Efficacy and Safety of Low Dose Rituximab Combined With Cyclosporine in the Treatment of Idiopathic Membranous Nephropathy
Brief Title: Efficacy of Rituximab Combined With Cyclosporine in the Treatment of Idiopathic Membranous Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wenhu Liu, Professor Wenhu Liu, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-P2-250-01
Record Dates: First submitted 2022-12-18; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental): Patients received rituximab 100 and 500 mg of intravenous medication on days 1 and 2, respectively. If proteinuria was reduced from baseline by no more than 25% at 3 months, cyclosporine was administered. In addition, CD19+ B-cell count was monitored every 3 months, and another rituximab 100 and 500 mg will be administered if CD19+ B-cell count >5 cells/mL.
  Interventions: Drug: Rituximab
- Modified Ponticelli regimen (Active Comparator): Patients received corticosteroids at months 1, 3, and 5 (methylprednisolone 0.5 g at days 1, 2, and 3, then prednisone 0.5 mg/kg/d from day-4 to day-30). At months 2, 4, and 6, patients received cyclophosphamide adjusted for age and renal function (1.0-2.0 mg/kg/day for 30 days, maximum dose 100 mg/d).
  Interventions: Drug: Modified Ponticelli regimen

INTERVENTIONS:
Drug: Rituximab — Rituximab combined with or without cyclosporine
  Arms: Rituximab
Drug: Modified Ponticelli regimen — Corticosteroid and cyclophosphamide
  Arms: Modified Ponticelli regimen

SUMMARY:
Idiopathic membranous nephropathy (IMN) is one of the common types of primary glomerular diseases and the most common cause of nephrotic syndrome in adults.

Poticelli regimen is the classic treatment, but cyclophosphamide has many toxic side effects. The period of glucocorticoid therapy is relatively long, and the adverse reactions caused by glucocorticoid therapy cannot be ignored. For patients who are unwilling to receive glucocorticoids and cyclophosphanide or who have treatment contraindications, cyclosporine can be used, mainly cyclosporine and tacrolimus, with the rapid overall effect but a high short-term relapse rate. In recent years, rituximab therapy has become a first-line treatment, with a high remission rate, and few side effects, but expensive. In terms of efficacy alone, the above regimen did not exceed Poticelli regimen. However, the toxic side effects of rituximab, cyclosporine may be lower than that of Poticelli regimen. Based on the preliminary experiment, this study explored a new treatment plan: low-dose rituximab combined with cyclosporine in the treatment of IMN, the efficacy is not inferior to Poticelli regimen, but the side effects are significantly reduced. The result will provide a good choice for IMN patients.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-70 years; serum albumin level <30 g/L;
2. estimated glomerular filtration rate (eGFR according to the CKD-EPI formula) ≥60 mL/min per 1.73 m2;
3. patients with a moderate risk of IMN and decline <50% in proteinuria despite blockade of the renin-angiotensin system 3 months before randomization;
4. patients at high risk or very high risk of IMN.

Exclusion Criteria:

1. secondary causes of MN;
2. being pregnant or breastfeeding;
3. uncontrollable active infectious disease;
4. immunosuppressive treatment in the preceding 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-12-04 (Estimated); Study Completion 2023-12-04 (Estimated)

PRIMARY OUTCOMES:
remission of nehprotic syndrome | 12 months
  The primary clinical outcome was a composite outcome with complete remission or partial remission of nehprotic syndrome at 12 months. Complete remission was defined as a reduction of proteinuria to ≤ 0.3 g/24 h plus stable kidney function (eGFR ≥45 mL/min per 1.73 m2). Partial remission was defined as a reduction of proteinuria of ≥ 50% from baseline, and <3.5 g/24 h plus stable renal function (eGFR ≥45 mL/min per 1.73 m2).

SECONDARY OUTCOMES:
Complete remission of nehprotic syndrome | 12 months
  Complete remission was defined as a reduction of proteinuria to ≤ 0.3 g/24 h plus stable kidney function (eGFR ≥45 mL/min per 1.73 m2).
adverse events | 12 months
  The prevalence of adverse events including infections, hyperglycemia etc will be recored.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China